CLINICAL TRIAL: NCT06921525
Title: Comparing Efficacy of Tea Tree Oil Versus Topical Azithromycin in Treating Dry Eye Disease Associated With Meibomian Gland Dysfunction: A Focus on Tear Interleukin Level
Brief Title: Comparing Efficacy of Tea Tree Oil Versus Topical Azithromycin in Treating Dry Eye
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ehab Mohamed Elsayed Mohamed Saad (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTO vs Azithromycine in MGD; Rewan Hassan Hamid Mohamoud (Other Grant/Funding Number: Demonstrator of Aharm canadian university); Dalia Refat El-Afify (Other Grant/Funding Number: Assistant professor of Clinical pharmacy Faculty of Pharmacy - Tanta University); Tamer Ibrahim Abdelhalim (Other Grant/Funding Number: Assistant professor of Ophthalmology Faculty of Medicine -Tanta University); Fedaa Abd Elmonem Kotkata (Other Grant/Funding Number: Lecturer of Clinical Pharmacy Faculty of Pharmacy - Tanta University)
Record Dates: First submitted 2025-03-23; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Azithromycin group) (Active Comparator): Group A (Azithromycin group): 22 patients who will receive topical azithromycin applied twice daily, along with preservative-free lubricant eye drops five times daily for 4 weeks.
  Interventions: Drug: Azithromycin Ophthalmic Solution
- Group B (Tea Tree Oil group) (Active Comparator): Group B (Tea Tree Oil group): 22 patients who will receive topical tea tree oil applied twice daily, along with preservative-free lubricant eye drops five times daily for 4 weeks.
  Interventions: Drug: Tea Tree Oil Topical Application Oil

INTERVENTIONS:
Drug: Tea Tree Oil Topical Application Oil — Tea tree oil (TTO), derived from the leaves of Melaleuca alternifolia,
  Arms: Group B (Tea Tree Oil group)
Drug: Azithromycin Ophthalmic Solution — Azithromycin has demonstrated efficacy in improving meibomian gland function and reducing inflammation and improving symptoms of dryness of the eye
  Arms: Group A (Azithromycin group)

SUMMARY:
This study aims to compare the effects of azithromycin and tea tree oil on the clinical outcomes and inflammatory profile of patients with MGD-associated DED. By focusing on changes in tear IL-8 and IL-17 levels, the study seeks to provide insights into the differential mechanisms of these two treatments and their potential in addressing inflammation-driven DED.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a multifactorial condition affecting the ocular surface, characterized by the loss of tear film homeostasis, resulting in discomfort, visual disturbances, and tear film instability . The prevalence of DED is significant, impacting approximately 5%-50% of the global population, with variability influenced by geographic location, age, and environmental factors . The condition not only affects the quality of life but also poses a substantial economic burden due to increased healthcare utilization and reduced productivity .

A hallmark of DED is its complex pathophysiology, which involves a vicious cycle of tear film instability, hyperosmolarity, and chronic inflammation of the ocular surface. Recent advances underscore the critical interplay between these factors and their contribution to symptomatology . Pro-inflammatory cytokines, such as interleukin-8 (IL-8) and interleukin-17 (IL-17), have emerged as key mediators of ocular surface inflammation, amplifying the recruitment of neutrophils and T-helper 17 cells, respectively .

Among the various etiologies of DED, meibomian gland dysfunction (MGD) is recognized as a leading cause. MGD results from abnormalities in the secretion of meibum, a lipid essential for stabilizing the tear film and preventing evaporation . Dysregulation of the lipid layer exacerbates evaporative dry eye and promotes a pro-inflammatory microenvironment, further destabilizing the tear film.

Conventional therapeutic approaches to MGD, such as warm compresses and eyelid hygiene, aim to restore gland function and relieve symptoms. In addition, topical antibiotics, particularly azithromycin, are commonly employed due to their dual antimicrobial and anti-inflammatory properties . Azithromycin has demonstrated efficacy in improving meibomian gland function and reducing inflammation and improving symptoms of dryness of the eye .

Emerging treatments for MGD have focused on addressing the underlying inflammatory and microbial components. Tea tree oil (TTO), derived from the leaves of Melaleuca alternifolia, has garnered attention due to its antimicrobial, anti-inflammatory, and demodicidal properties . TTO has demonstrated efficacy in eradicating Demodex mites, microscopic parasites frequently associated with MGD and DED . Despite these promising effects, its impact on tear cytokine modulation remains an area of active investigation .

Preclinical and clinical studies have begun to elucidate the mechanisms by which TTO exerts its effects. For instance, TTO has been shown to inhibit pro-inflammatory pathways, reduce oxidative stress, and enhance epithelial barrier integrity . These findings suggest a broader therapeutic role for TTO in addressing not only MGD but also other ocular surface diseases characterized by inflammation and microbial dysbiosis .

Despite its potential, challenges remain in the widespread adoption of TTO for MGD. Patient tolerability, particularly regarding ocular irritation, is a critical consideration. Additionally, the lack of large-scale, randomized controlled trials limits the generalizability of existing findings .

In conclusion, while conventional therapies for MGD have been effective, emerging treatments such as TTO offer a promising alternative, particularly in addressing inflammation and microbial factors. Understanding the interplay between TTO, cytokines like IL-8 and IL-17, and the ocular surface could pave the way for novel therapeutic paradigms, ultimately improving outcomes for patients with DED and MGD .

ELIGIBILITY:
Inclusion Criteria:

* Tear Break-Up Time (TBUT) ≤10 seconds.
* Ocular Surface Disease Index (OSDI) score ≥20.
* Willingness to comply with study requirements and provide informed consent.

Exclusion Criteria:

* History of ocular surgery or trauma within the past 6 months.
* Use of systemic or topical anti-inflammatory medications within 4 weeks prior to enrollment.
* Known hypersensitivity to azithromycin or tea tree oil.
* Presence of other ocular surface diseases unrelated to MGD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in IL-8 and IL-17 levels . | after 4 weeks of treatment

SECONDARY OUTCOMES:
Change in clinical parameters (TBUT, OSDI, DEQS, Schirmer test). | after 4 weeks of treatment
  Change in the parameters TBUT "Tear breakup time'', OSDI ''Ocular Surface Disease Index'', DEQS ''Dry Eye-Related Quality-of-Life Score'' and Schirmer test.
  TBUT (from less than 5 to more than 10 seconds). OSDI (from 0 to 100 points) where patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time" a final score is calculated which ranges from 0 to 100 with scores and based on their OSDI scores, patients can be categorized as having a normal ocular surface (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) ocular surface disease.
  DEQS (from 0 to 100 points) which is a questionnaire and it was calculated using the following formula: (sum of the degree scores for all questions answered) × 25/(total number of questions answered), with higher scores indicating increased severity of DED symptoms and a greater impact on daily life.
  Schirmer test (from 0 to 15 mm).
Change in meibomian gland function grading (from 0 to 4) | after 4 weeks of treatment
Change in parameter OSDI (ocular surface disease index) from 0 to 100 points. | after 4 weeks of treatment
  OSDI (from 0 to 100 points) where patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time" a final score is calculated which ranges from 0 to 100 with scores and based on their OSDI scores, patients can be categorized as having a normal ocular surface (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) ocular surface disease.
Change in the parameter DEQS (Dry Eye-Related Quality-of-Life Score) from 0 to 100 points. | after 4 weeks of treatment
  DEQS (from 0 to 100 points) which is a questionnaire and it was calculated using the following formula: (sum of the degree scores for all questions answered) × 25/(total number of questions answered), with higher scores indicating increased severity of DED symptoms and a greater impact on daily life.
Change in the parameter Schirmer test (from 0 to 15 mm). | after 4 weeks of treatment
  Change in the parameter Schirmer test (from 0 to 15 mm) as Schirmer test results are interpreted as follows: 0 to 5 mm: extremely dry eyes. 5 to 10 mm: moderately dry eyes. 10 to 15 mm: possible dry eyes.